CLINICAL TRIAL: NCT00121225
Title: A Phase II Study of Vorinostat in Patients With Advanced Melanoma
Brief Title: Vorinostat in Treating Patients With Metastatic or Unresectable Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00099; PHL-040 (Other Grant/Funding Number: N01CM62203); CDR0000436851 (Other Grant/Funding Number: N01CM62203); N01CM62203 (NIH)
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Ciliary Body and Choroid Melanoma, Medium/Large Size; Extraocular Extension Melanoma; Iris Melanoma; Uveal Melanoma; Recurrent Intraocular Melanoma; Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients will receive vorinostat by mouth once a day for 4 weeks. Treatment may repeat every 4 weeks for as long as benefit is shown. Patients will be evaluated for 4 weeks and every 3 months thereafter.
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — Patients will receive vorinostat by mouth once a day for 4 weeks. Treatment may repeat every 4 weeks for as long as benefit is shown. Patients will be evaluated for 4 weeks and every 3 months thereafter.
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza

SUMMARY:
This phase II trial is studying how well vorinostat works in treating patients with metastatic or unresectable melanoma. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the objective response rate in patients with metastatic or unresectable melanoma treated with vorinostat.

SECONDARY OBJECTIVES:

I. Determine time to progression in patients treated with this drug. II. Determine the utility of HP1 and/or macro H2A nuclear foci as biomarkers of response in patients treated with this drug.

III. Correlate the presence of 72R or 72P variant p53 polymorphisms with response and time to progression in patients treated with this drug.

IV. Determine gene expression profiles that may predict response to this drug and gene expression changes that occur after treatment with this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral vorinostat once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed melanoma that is metastatic/unresectable
* Residual, recurrent, or metastatic disease by radiographic examination. Measurable disease (at least 1 lesion in at least 1 dimension (longest diameter) as >20mm with conventional techniques or >10mm with spiral CT scan, within 4 weeks prior to registration
* No prior therapy or 1 prior treatment (cytokine/chemotherapy/combination) for metastatic disease allowed. Patients should not take valproic acid, another histone deacetylase inhibitor, for at least 2 weeks prior to enrollment. At least 4 weeks from prior therapy to be eligible or 6 weeks if last regimen included BCNU or mitomycin C
* Age>=18 years
* Life expectancy >=3 months.
* ECOG<2 (Karnofsky ≥60%)
* Leukocytes >3,000/mcL
* Absolute neutrophil count >1,500/mcL
* Platelets >100,000/mcL
* Total bilirubin within institutional limits
* AST/ALT≤2.5Xinstitutional ULN
* Creatinine within institutional limits OR creatinine clearance >60mL/min/1.73 m2 if creatinine levels above institutional limits
* Eligibility of patients taking medications with potential to affect activity/PK of Vorinostat will be determined by PI
* Must not use concomitant steroids except topical/inhaled use
* Vorinostat effects on developing human fetus are unknown. Women of childbearing potential (WOCBP) and sexually active males must agree to use accepted/effective contraception method prior to study entry and for duration of the study
* Ability to understand/willingness to sign written informed consent
* Must have paraffin block of tumor tissue available for future studies

Exclusion Criteria:

* Chemotherapy/radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering study
* May not be receiving any other investigational agents
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical/biologic composition to Vorinostat
* Uncontrolled intercurrent illness including but not limited to ongoing/active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women excluded because Vorinostat is a HDAC inhibitor agent with potential for teratogenic or abortifacient effects
* HIV-positive patients receiving combination antiretroviral therapy are ineligible because of potential for PK interactions with Vorinostat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Balzer-Haas, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (5):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Rockledge, Pennsylvania
- Canada (3):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Result] Haas NB, Quirt I, Hotte S, McWhirter E, Polintan R, Litwin S, Adams PD, McBryan T, Wang L, Martin LP, vonMehren M, Alpaugh RK, Zweibel J, Oza A. Phase II trial of vorinostat in advanced melanoma. Invest New Drugs. 2014 Jun;32(3):526-34. doi: 10.1007/s10637-014-0066-9. Epub 2014 Jan 25. PMID 24464266

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Vorinostat: Patients will receive vorinostat by mouth once a day for 4 weeks. Treatment may repeat every 4 weeks for as long as benefit is shown. Patients will be evaluated for 4 weeks and every 3 months thereafter.
  vorinostat
Period: Overall Study
Arm/Group | Arm 1 Vorinostat
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients will receive vorinostat by mouth once a day for 4 weeks. Treatment may repeat every 4 weeks for as long as benefit is shown. Patients will be evaluated for 4 weeks and every 3 months thereafter.
  vorinostat
Arm/Group | Arm I
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 61 [38 to 89]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 13
  Canada | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Assessed by Response Evaluation Criteria for Solid Tumors (RECIST)
Description: Per Response Evaluation Criteria in Solid Tumours Criteria (RECIST v1.0) for target lesions and are assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least 30% decrease in sum of longest diameter of target lesions; Objective Response (OR) = CR+ PR.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 32
participants | 2

2. Secondary Outcome: Time to Progression Assessed by RECIST
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 Vorinostat
Number analyzed (Participants) | 32
months | 4 [1.8 to 4]

3. Secondary Outcome: Difference in HP1 and MacroH2A Nuclear Foci Expression Between Progressive Minus Stable Disease Outcomes
Description: Macro H2A and HP1 expression levels were compared through analysis of log fold changes in antibody expression in a multivariate general linear model between progressive disease and stable disease outcomes.
Time Frame: Baseline and day 15
Population: Patient 32 had pre-treatment punch biopsy that was inadequate for testing, thus was not included in this measurement
Measure: Mean (Standard Error); unit: log fold change
Arm/Group | Arm 1 Vorinostat
Number analyzed (Participants) | 31
log fold change
  MacroH2A1.1 | 0.149 (0.364)
  MacroH2A1.2 | -0.748 (0.466)
  HP1 | -0.077 (0.395)

4. Secondary Outcome: Number of Patients With p53 Allelic Variations (72R or 72P)
Description: Participants were assessed for p53 allelic variation at baseline
Time Frame: Baseline
Population: Participant 32 had a pre-treatment punch biopsy that was not adequate for testing
Measure: Number; unit: participants
Arm/Group | Arm 1 Vorinostat
Number analyzed (Participants) | 31
participants
  Wild Type | 20
  Mutant | 11

5. Secondary Outcome: Comparison of VEGF Serum Levels to Response to Vorinostat
Description: Blood specimens were collected from participants on Day 1 Cycle 1 prior to treatment (baseline), Day 1 3-4 hours following Vorinostat ingestion, Day 8 and Day 15. VEGF serum concentrations were detected using the Luminex multiplexed assay, where the median fluorescence intensity results were analyzed by a weighted five-parameter logistic method. The values were averaged across all time points per participant.
Time Frame: Baseline, Day 1, Day 8 and Day 15
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Arm 1 Vorinostat
Number analyzed (Participants) | 32
pg | 203 (0.029)
Statistical Analysis 1: Comparison: Arm 1 Vorinostat; Test type: Superiority; p = 0.029, Fisher Exact

ADVERSE EVENTS:
Description: Indicates events were collected by systematic assessment and are reported regardless of attribution to agent.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 9/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=32)
Dry mouth (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Platelet count decreased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1 — unrelated to study drug
Hyperglycemia (Metabolism and nutrition disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=32)
Fatigue (General disorders) | 28
Hyperglycemia (Metabolism and nutrition disorders) | 24
Anemia (Blood and lymphatic system disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less